CLINICAL TRIAL: NCT00281151
Title: Center for Reducing Asthma Disparities - Meharry/Vanderbilt Centers
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University School of Medicine (Other); Meharry Medical College (Other)
Responsible Party: Principal Investigator, James Sheller, Professor of Medicine, Vanderbilt University
Other Study IDs: 1198; U01HL072431 (NIH); U01HL072471 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2009-02

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the mechanisms underlying the disparities in asthma and to improve asthma care in pregnant women, a targeted group at high risk for asthma-specific maternal and perinatal complications.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic condition affecting over 14 million Americans. Data indicate that rates of asthma are higher in certain populations. In fact, African Americans and Hispanics from the Northeast are twice as likely to die from asthma as whites. African Americans are four times as likely to be hospitalized for asthma and are five times more likely than whites to seek care for asthma at an emergency department. Reasons for these higher rates are not certain, and most likely result from an interaction of risk factors such as environmental exposures, genetic predisposition, access to appropriate medical care, socioeconomic status, and cultural health practices. The National Heart, Lung, and Blood Institute (NHLBI) supports a variety of activities to address the pressing public health problems posed by asthma. However, progress in reducing disparities has been disappointingly slow. Separate, independent research projects have generated important clues for understanding the nature and scope of the problem, but a more coordinated, interdisciplinary, and comprehensive approach to research is needed. By fostering partnerships among minority medical centers, research intensive institutions, and the communities in which asthma patients live, cooperative research centers can help increase the capacity to improve health outcomes among minority and economically disadvantaged populations.

DESIGN NARRATIVE:

This study will comprise three groups: pregnant women with asthma, children requiring intensive care unit (ICU) admission for asthma, and asthmatics requiring emergency care. In one part of the study, researchers will randomly assign pregnant women with asthma of African American or Hispanic race/ethnicity to one of two culturally sensitive asthma education and smoking cessation programs. At the same time, investigators will examine asthma-related morbidity in a large cohort of pregnant asthmatic women utilizing administrative data and vital records. Perceptions of asthma severity and ways to describe it appear to differ in African Americans compared to whites. Therfore, asthmatic patients attending the emergency room, along with their families, will be invited to participate in a focus group to validate a culturally sensitive instrument to allow improved descriptors of asthma severity for African Americans. Estimates by the patients of asthma severity will be matched to objective measure, and compared with those of whites. This methodology will then be used to extend the hypothesis to children admitted with severe asthma to the region's only pediatric ICU. In the pediatric ICU, the admission rates and outcomes will be associated with the potentially important genetic variations in the beta 2 adrenergic receptor (BADR2). Using parents and non-affected siblings as case controls, a novel computational method will test for gene-gene interactions that explain a genetic basis for asthma disparities in severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with asthma
* Children requiring intensive care unit (ICU) admission for asthma
* Asthmatics requiring emergency care.

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll pregnant women with asthma, children requiring intensive care unit (ICU) admission for asthma, and asthmatics requiring emergency care.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2002-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Asthma related maternal/fetal morbidities and asthma control | Measured between two and six weeks following delivery

CONTACTS AND LOCATIONS:
Overall Officials: James R. Sheller, Principal Investigator — Vanderbilt University Medical Center; John J. Murray, Principal Investigator — Meharry Medical School
Locations (2):
- United States (2):
  - Meharry Medical School, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Talbot TR, Hartert TV, Mitchel E, Halasa NB, Arbogast PG, Poehling KA, Schaffner W, Craig AS, Griffin MR. Asthma as a risk factor for invasive pneumococcal disease. N Engl J Med. 2005 May 19;352(20):2082-90. doi: 10.1056/NEJMoa044113. PMID 15901861
- [Background] Whalen U, Griffin MR, Shintani A, Mitchel E, Cruz-Gervis R, Forbes BL, Hartert TV. Smoking rates among pregnant women in Tennessee, 1990-2001. Prev Med. 2006 Sep;43(3):196-9. doi: 10.1016/j.ypmed.2006.04.021. Epub 2006 Jun 15. PMID 16780937
- [Background] Enriquez R, Wu P, Griffin MR, Gebretsadik T, Shintani A, Mitchel E, Carroll KN, Hartert TV. Cessation of asthma medication in early pregnancy. Am J Obstet Gynecol. 2006 Jul;195(1):149-53. doi: 10.1016/j.ajog.2006.01.065. Epub 2006 May 2. PMID 16631099
- [Background] Carroll KN, Griffin MR, Gebretsadik T, Shintani A, Mitchel E, Hartert TV. Racial differences in asthma morbidity during pregnancy. Obstet Gynecol. 2005 Jul;106(1):66-72. doi: 10.1097/01.AOG.0000164471.87157.4c. PMID 15994619
- [Background] Hartert TV, Neuzil KM, Shintani AK, Mitchel EF Jr, Snowden MS, Wood LB, Dittus RS, Griffin MR. Maternal morbidity and perinatal outcomes among pregnant women with respiratory hospitalizations during influenza season. Am J Obstet Gynecol. 2003 Dec;189(6):1705-12. doi: 10.1016/s0002-9378(03)00857-3. PMID 14710102
- [Background] Venarske DL, Busse WW, Griffin MR, Gebretsadik T, Shintani AK, Minton PA, Peebles RS, Hamilton R, Weisshaar E, Vrtis R, Higgins SB, Hartert TV. The relationship of rhinovirus-associated asthma hospitalizations with inhaled corticosteroids and smoking. J Infect Dis. 2006 Jun 1;193(11):1536-43. doi: 10.1086/503809. Epub 2006 Apr 27. PMID 16652282